CLINICAL TRIAL: NCT01779739
Title: Evaluating Sexual Function After Vaginal Repair With Perineorrhaphy
Acronym: FaVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00037135; NCT03333811 (obsolete NCT alias)
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Sexual Function
Keywords: vaginal prolapse; sexual function; sexual dysfunction; prolapse surgery
MeSH Terms: conditions — Uterine Prolapse; Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No perineorrhaphy (No Intervention): Subjects will not have a perineorrhaphy procedure added to the vaginal prolapse repair
- Perineorrhaphy (Active Comparator): Subjects will have a perineorrhaphy added to the vaginal repair of prolapse
  Interventions: Procedure: Perineorrhaphy

INTERVENTIONS:
Procedure: Perineorrhaphy — Procedure to build up the vaginal opening
  Arms: Perineorrhaphy

SUMMARY:
This is a single center, double-blind, randomized controlled trial evaluating the change in sexual function in women undergoing vaginal repair for pelvic organ prolapse. Participants will be sexually active women who agree to randomization to having perineorrhaphy added to or excluded from their surgical repair. We hypothesize that sexual function will improve more significantly in women undergoing vaginal repair with perineorrhaphy.

ELIGIBILITY:
Inclusion Criteria:

* sexually active
* genital hiatus measured between 4 and 6 centimeters
* desires sexual function
* undergoing vaginal repair with native tissues
* agrees to use vaginal estrogen for 12 months after surgery

Exclusion Criteria:

* genital hiatus > 6 cm
* planned obliterative procedure
* perineal body length <0.5cm
* disrupted external anal sphincter

Ages: 19 Years to 105 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-07; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in sexual function as measured by validated questionnaire | 6 months and 12 months after surgery
  Validated questionnaires will be administered prior to surgery, as well as at intervals after surgery.

SECONDARY OUTCOMES:
Prolapse recurrence | 6 months, 12 months
  A composite outcome score to define success of prolapse surgery will be applied to subjects at 6 and 12 months specifically looking for return of prolapse symptoms, anatomic recurrence, and need for retreatment

CONTACTS AND LOCATIONS:
Overall Officials: Candace Y Parker-Autry, MD, Study Director — Wake Forest; Holly E Richter, PhD, MD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina